CLINICAL TRIAL: NCT00070265
Title: A Multi-Institutional Phase II Trial Of Neoadjuvant Capecitabine (XELODA) And Oxaliplatin (ELOXATIN) For Resectable Colorectal Metastases In The Liver
Brief Title: Neoadjuvant and Adjuvant Capecitabine and Oxaliplatin in Treating Patients With Resectable Liver Metastases Secondary to Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02722; MDA-ID-02636; N01CM17003 (NIH); CDR0000331853 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Liver Metastases; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine

ARMS (1):
- Treatment (oxaliplatin, capecitabine, and surgery) (Experimental): Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Surgery: Four to six weeks after the completion of chemotherapy, patients undergo surgical resection of the tumor.
  Adjuvant chemotherapy: Patients with satisfactory response to therapy receive 4 additional courses of oxaliplatin and capecitabine after surgery.
  Interventions: Drug: oxaliplatin; Drug: capecitabine; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as capecitabine and oxaliplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Giving capecitabine and oxaliplatin before surgery may shrink the tumor so that it can be removed. Giving capecitabine and oxaliplatin after surgery may kill any remaining tumor cells. This phase II trial is studying how well capecitabine and oxaliplatin work when given before and after surgery in treating patients with resectable liver metastases that is secondary to colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy and toxicity of neoadjuvant and adjuvant capecitabine and oxaliplatin in patients with resectable liver metastases secondary to colorectal cancer who are undergoing surgery.

II. Determine the rates of R0 resection in patients treated with this regimen before surgery.

SECONDARY OBJECTIVES:

I. Determine the response rate in patients treated with this regimen. II. Determine the resectability in the subsets of patients defined as resectable preoperatively and treated with this regimen.

III. Determine improvement in survival associated with downstaging based on metastatic colorectal prognostic score in patients treated with this regimen.

IV. Determine the disease-free and overall survival of patients treated with this regimen.

V. Correlate drug-specific biomarkers with clinical response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Surgery: Four to six weeks after the completion of chemotherapy, patients undergo surgical resection of the tumor.

Adjuvant chemotherapy: Patients with satisfactory response to therapy receive 4 additional courses of oxaliplatin and capecitabine after surgery.

Patients are followed at 4-6 weeks after surgery, every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 80 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hepatic colorectal metastasis by percutaneous hepatic biopsy

  * Imaging evidence of liver metastasis by CT helical scan
* Resectable disease, as determined by a surgeon with hepatic surgery expertise (at least 10 resections performed per year)

  * Resectable, defined as a sparing of 2 adjacent liver segments with adequate vascular inflow and outflow and hepatic remnant volume
  * Minor resections (less than a hemihepatectomy) or major resections (hemihepatectomy or extended hepatectomy) allowed
  * Bilobar resection allowed, including atypical resections
* No evidence of extrahepatic disease by chest x-ray or CT scan of the chest, abdomen, and pelvis
* Performance status - Zubrod 0-1
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 2 mg/dL
* AST and ALT no greater than 300 IU/L
* No preexisting chronic hepatic disease (e.g., chronic active hepatitis or cirrhosis) that would preclude surgical resection of metastases
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except completely resected nonmelanoma skin cancer or carcinoma in situ of the cervix
* No preexisting grade 2 or greater peripheral neuropathy
* No concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent biologic therapy
* No concurrent sargramostim (GM-CSF)
* More than 6 months since prior adjuvant fluorouracil-based chemotherapy
* No prior chemotherapy for liver metastasis
* No prior oxaliplatin for colorectal cancer
* No prior or concurrent hepatic artery infusion chemotherapy for metastatic disease
* No prior or concurrent radiotherapy for metastatic disease
* No prior or concurrent radiofrequency ablation for metastatic disease
* No prior or concurrent cryotherapy/other ablative techniques for metastatic disease
* No other concurrent investigational therapy
* No concurrent oral anticoagulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-08; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Rate of complete resection (R0 resection) | Up to 5 years
  The design of Thall and Simon will be used.

SECONDARY OUTCOMES:
Response rate assessed using RECIST criteria | Up to 5 years
Resectability in the subsets defined as resectable preoperatively | Up to 5 years
Improvement in survival associated with downstaging based on metastatic colorectal prognostic score | Up to 5 years
Disease-free survival | Up to 5 years
Overall survival | Up to 5 years
Positron emission tomography response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Vauthey, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas, Houston, Texas, United States